CLINICAL TRIAL: NCT02407444
Title: A Comparison of Two Physiotherapy Treatment Protocols, With and Without Cycling Training , in Elderly Patients With Hip Fractures at Their Subacute Stage Following Surgery
Brief Title: Treatment Efficacy of Leg Cycling as Part of Physiotherapy Treatment in Elderly Patients With Hip Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Beit-Rivka Geriatric Rehabilitation Hospital (Unknown)
Responsible Party: Principal Investigator, AVITAL HERSHKOVITZ, MD, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rmc150495ctil
Record Dates: First submitted 2015-03-19; First posted 2015-04-03 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Hip Fractures
Keywords: Proximal hip fracture; Elderly patients; Physiotherapy; Leg cycling ergometer
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapy treatment & leg cycling (Experimental): This group will receive conventional physiotherapy treatments, each session will last 30 minutes. Treatments include muscles strength exercises for upper and lower extremities, static and dynamic balance training in standing ,pain relief techniques and functional training (including transfers, sit to stand, walking and climbing stairs). The treatment program shall be consistent with the patient's problems and the degree of difficulty will rise depending on progress.
  In addition this group will have cycling training with leg cycle ergometer for 20 minutes.
  This treatment protocol will last for three weeks, five days a week, 50 minutes each session per day.
  Interventions: Other: Physiotherapy treatment & leg cycling
- Physiotherapy treatment & music listening (Active Comparator): This group will receive conventional physiotherapy treatments, each session will last 30 minutes .Treatments include muscles strength exercises for upper and lower extremities, static and dynamic balance training in standing ,pain relief techniques and functional training (including transfers, sit to stand, walking and climbing stairs). The treatment program shall be consistent with the patient's problems and the degree of difficulty will rise depending on progress.
  In addition this group will listen to music (while sitting on a chair) for 20 minutes.This treatment protocol will last for three weeks, five days a week, 50 minutes each session per day.
  Interventions: Other: Physiotherapy treatment & music listening

INTERVENTIONS:
Other: Physiotherapy treatment & leg cycling — All patients receive comprehensive care as part of routine rehabilitation program : individual physical therapy treatment, gym's training and balance training in virtual reality, occupational therapy treatment, strengthening and range of motion exercises as a group.
  In addition each patient in this group will train with stationary leg cycle ergometer for 20 minutes under physical therapist's supervision . Cycling exercise intensity subjectively determined by the patient using RPE Borg scale . Maximal intensity level determined as 14 in Borg scale.
  Arms: Physiotherapy treatment & leg cycling
Other: Physiotherapy treatment & music listening — All patients receive comprehensive care as part of routine rehabilitation program : individual physical therapy treatment, gym's training and balance training in virtual reality, occupational therapy treatment, strengthening and range of motion exercises as a group.
  In addition each patient in this group will listen to music with earphone for 20 minutes while sitting under physical therapist supervision.
  Overall treatment session will last 50 minutes.
  Arms: Physiotherapy treatment & music listening

SUMMARY:
This study aims to evaluate whether a combination of cycling training as part of physiotherapy treatment will contribute more than conventional physiotherapy treatment for elderly patients after hip fracture surgery in their subacute phase of rehabilitation.

DETAILED DESCRIPTION:
Adults who have experienced a fall, followed by proximal hip fracture that required surgery, suffer from specific problems that interrupt the rehabilitation period in their subacute phase.

Various modes of treatment available as part of the physical rehabilitation but there is not enough data in the literature regarding the contribution of cycling training with leg cycle ergometer as part of conventional physiotherapy treatment in elderly patients after hip fracture surgery.

This study evaluates whether the additional cycling to physiotherapy treatment will improve the functional ability, the balance performance while standing, hip muscle strength and pain level in those patients.

ELIGIBILITY:
Inclusion Criteria:

* Proximal hip fracture with full or partial weight bearing indication.
* Surgical fixation ( nailing or total hip replacement or hemiarthroplasty)
* Pre-morbid function: walking independently or under supervision with or without assistance aid
* Cognitive function: Mini-mental state examination score above 21

Exclusion Criteria:

* Pathological hip fracture.
* Unstable heart or pulmonary disease.
* Presence of other fractures as a result of the current fall.
* Neurological comorbidities ( CVA, Parkinson, MS ).
* Entering the rehabilitation center more than three weeks after hip surgery

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-05 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
FIM ( functional independence measure) | baseline-at the first day of intervention
  Provides a uniform system of measurement for disability, it measures the level of patient's disability and indicates how much assistance is required for the individual to carry out activities of daily living. It contains 18 items composed of 13 motor tasks and 5 cognitive tasks. Tasks are rated on 7 point ordinal scale that ranges from total assistance to complete independence. Score range from 18 (lowest) to 126 (highest) indicating level of function.
Static balance test and weight bearing distribution while standing | baseline-at the first day of intervention
  The balance and weight bearing distribution parameters will be evaluated by posturographic device . This system assesses pressure fluctuations produced by the heels and toes of a subject standing on four separate platforms two for each foot and their respective halves. The pressure plates emit electronic signals which are digitized and processed by the posturographic device software to yield a set of unique parameters. Calculated results based on these parameters, which are statistically and functionally independent, reflect the interactions of the various neuro-physiological and neuro-anatomic subsystems involved in balance control.
Muscle strength | baseline-at the first day of intervention
  Quadriceps strength and hand grip will be assessed by hand held dynamometer. This is a quantitative and objective method for assessment of muscular strength. Scored using force production in kilograms.
Pain intensity (measured with VAS) | baseline-at the first day of intervention
  Subjective pain intensity will be measured with VAS which is an 11 point scale from 0-10, "0" indicates no pain and "10" indicates the most intense pain imaginable. The patient select the value that is most in line with the intensity of pain that he experienced in the last 24 hours.
Change from baseline in FIM at 2 weeks | Second week of intervention
  Provides a uniform system of measurement for disability, it measures the level of patient's disability and indicates how much assistance is required for the individual to carry out activities of daily living. It contains 18 items composed of 13 motor tasks and 5 cognitive tasks. Tasks are rated on 7 point ordinal scale that ranges from total assistance to complete independence. Score range from 18 (lowest) to 126 (highest) indicating level of function.
Change from baseline in FIM at 3 weeks | End of intervention at third week
  Provides a uniform system of measurement for disability, it measures the level of patient's disability and indicates how much assistance is required for the individual to carry out activities of daily living. It contains 18 items composed of 13 motor tasks and 5 cognitive tasks. Tasks are rated on 7 point ordinal scale that ranges from total assistance to complete independence. Score range from 18 (lowest) to 126 (highest) indicating level of function.
Change from baseline in static balance test and weight bearing distribution while standing at 2 weeks | Second week of intervention
  The balance and weight bearing distribution parameters will be evaluated by posturographic device . This system assesses pressure fluctuations produced by the heels and toes of a subject standing on four separate platforms two for each foot and their respective halves. The pressure plates emit electronic signals which are digitized and processed by the posturographic device software to yield a set of unique parameters. Calculated results based on these parameters, which are statistically and functionally independent, reflect the interactions of the various neuro-physiological and neuro-anatomic subsystems involved in balance control.
Change from baseline in static balance test and weight bearing distribution while standing at 3 weeks | End of intervention at third week
  The balance and weight bearing distribution parameters will be evaluated by posturographic device . This system assesses pressure fluctuations produced by the heels and toes of a subject standing on four separate platforms two for each foot and their respective halves. The pressure plates emit electronic signals which are digitized and processed by the posturographic device software to yield a set of unique parameters. Calculated results based on these parameters, which are statistically and functionally independent, reflect the interactions of the various neuro-physiological and neuro-anatomic subsystems involved in balance control.
Change from baseline in muscle strength at 2 weeks | Second week of intervention
  Quadriceps strength and hand grip will be assessed by hand held dynamometer. This is a quantitative and objective method for assessment of muscular strength. Scored using force production in kilograms.
Change from baseline in muscle strength at 3 weeks | End of intervention at third week
  Quadriceps strength and hand grip will be assessed by hand held dynamometer. This is a quantitative and objective method for assessment of muscular strength. Scored using force production in kilograms.
Change from baseline in pain intensity at 2 weeks (measured with VAS) | Second week of intervention
  Subjective pain intensity will be measured with VAS which is an 11 point scale from 0-10, "0" indicates no pain and "10" indicates the most intense pain imaginable. The patient select the value that is most in line with the intensity of pain that he experienced in the last 24 hours.
Change from baseline in pain intensity at 3 weeks (measured with VAS) | End of intervention at third week
  Subjective pain intensity will be measured with VAS which is an 11 point scale from 0-10, "0" indicates no pain and "10" indicates the most intense pain imaginable. The patient select the value that is most in line with the intensity of pain that he experienced in the last 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Avital Hershkovitz, MD-PhD, Principal Investigator — Beit-Rivka Geriatric Rehabilitation Hospital; Youssef Ma Masharawi, PhD, Study Chair — Tel Aviv University
Locations (1):
- "Beit- Rivka" geriatric rehabilitation hospital, Petach Tiqva, Israel

REFERENCES:
- [Derived] Fairhall NJ, Dyer SM, Mak JC, Diong J, Kwok WS, Sherrington C. Interventions for improving mobility after hip fracture surgery in adults. Cochrane Database Syst Rev. 2022 Sep 7;9(9):CD001704. doi: 10.1002/14651858.CD001704.pub5. PMID 36070134